CLINICAL TRIAL: NCT00447980
Title: A Phase II/III Study of Encapsulated Human NTC-201 Cell Implants Releasing Ciliary Neurotrophic Factor (CNTF) for Participants With Retinitis Pigmentosa Using Visual Field Sensitivity as the Primary Outcome
Brief Title: A Study of Encapsulated Cell Technology (ECT) Implant for Participants With Early Stage Retinitis Pigmentosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurotech Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNTF 4
Record Dates: First submitted 2007-03-09; First posted 2007-03-15 (Estimated); Results first posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinitis Pigmentosa; eye disease; retinal disorder; CNTF
MeSH Terms: conditions — Retinitis Pigmentosa; Eye Diseases; Retinal Diseases | interventions — Ciliary Neurotrophic Factor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Dose (Experimental): NT-501 Low Dose Implant: encapsulated cell therapy that delivers ciliary neurotrophic factor to the retina
  Sham Implant in Fellow Eye
  Interventions: Drug: NT-501
- High Dose (Experimental): NT-501 High Dose Implant: encapsulated cell therapy that delivers ciliary neurotrophic factor to the retina
  Sham Implant in Fellow Eye
  Interventions: Drug: NT-501

INTERVENTIONS:
Drug: NT-501 — Low Dose
  Other Names: CNTF implant
  Arms: Low Dose
Drug: NT-501 — High Dose
  Other Names: CNTF implant
  Arms: High Dose

SUMMARY:
The purpose of this study is to look at the safety and effectiveness of CNTF implants on vision in persons with retinitis pigmentosa, Usher type II & III, and Choroideremia. This research is being done because there are no effective therapies for people with these retinal degenerations. They are genetic disorders that affect one's ability to see at night, and later cause tunnel vision and loss of central vision. Retinal degenerations affect the retina, a light sensitive layer of cells in the back of the eye. Slowly over time, these cells die and cause permanent loss of vision.

The implant is a small capsule that contains human retinal pigment epithelium cells. These cells have been given the ability to make CNTF and release it through the capsule membrane into the surrounding fluid. In this study, two different CNTF dose levels will be used: a high dose and a low dose in one eye, as well as a sham (or placebo) surgery in the other eye.

DETAILED DESCRIPTION:
This study will involve about 18 visits over 2½ years for specific tests of the participant's vision and health. These visits may include visual exams, blood draw for laboratory testing, brief medical history and exam, and occasionally a questionnaire (survey), in addition to the visit for the surgical procedures. The primary effectiveness outcome for this study will be a visual field score one year after the implant surgery. There will be about 12 centers participating in this study, and up to 60 people enrolled, across the US. Each participant joining the study who has completed initial screening will then be scheduled to have a brief surgical procedure performed on each eye, one of which will include a very small cell-filled implant. Follow-up visits for repeat assessments will be required regularly to determine if the implant being tested is safe and effective for use to treat retinitis pigmentosa (RP).

ELIGIBILITY:
Study inclusion / exclusion criteria:

Criteria for patients to qualify for the study include, but are not limited to:

* Over 18 years of age, and less than 65 years of age
* Diagnosis of retinitis pigmentosa, Usher Syndrome Type 2 or 3 or Choroideremia
* Visual acuity no worse than 20/63
* Experience with at least two full threshold Humphrey Visual Field 30-2 tests, one completed within the year prior to enrolling in this study

The following criteria will exclude patients from the study:

* Pregnant or lactating females, or females planning to become pregnant during the study or not using an acceptable method of contraception.
* Retinitis pigmentosa caused by a classic syndrome, including Usher Type I
* Other eye diseases including advanced cataract.
* Chronic systemic disease requiring continuous treatment with systemic steroids, immunosuppressive medications or insulin.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2007-01-22 (Actual); Primary Completion 2010-04-19 (Actual); Study Completion 2010-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Birch, MD, PhD, Principal Investigator — Retina Foundation of the Southwest
Locations (12):
- United States (12):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - University of Califoria, Davis, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - Bascom Palmer Eye Insitute, Miami, Florida
  - Kellogg Eye Center, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - NY University Medical Center, New York, New York
  - Casey Eye Institue, Portland, Oregon
  - The Hamilton Eye Institute, Memphis, Tennessee
  - Retina Foundation of Southwest, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - The University of Utah - John A. Moran Eye Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Birch DG, Weleber RG, Duncan JL, Jaffe GJ, Tao W; Ciliary Neurotrophic Factor Retinitis Pigmentosa Study Groups. Randomized trial of ciliary neurotrophic factor delivered by encapsulated cell intraocular implants for retinitis pigmentosa. Am J Ophthalmol. 2013 Aug;156(2):283-292.e1. doi: 10.1016/j.ajo.2013.03.021. Epub 2013 May 10. PMID 23668681
- [Derived] Kauper K, McGovern C, Sherman S, Heatherton P, Rapoza R, Stabila P, Dean B, Lee A, Borges S, Bouchard B, Tao W. Two-year intraocular delivery of ciliary neurotrophic factor by encapsulated cell technology implants in patients with chronic retinal degenerative diseases. Invest Ophthalmol Vis Sci. 2012 Nov 1;53(12):7484-91. doi: 10.1167/iovs.12-9970. PMID 23049090
- [Derived] Talcott KE, Ratnam K, Sundquist SM, Lucero AS, Lujan BJ, Tao W, Porco TC, Roorda A, Duncan JL. Longitudinal study of cone photoreceptors during retinal degeneration and in response to ciliary neurotrophic factor treatment. Invest Ophthalmol Vis Sci. 2011 Apr 6;52(5):2219-26. doi: 10.1167/iovs.10-6479. PMID 21087953

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 90 participants were screened and 73 were randomized to dose groups. 17 of 90 patients were screen failures and not associated (randomized) to either arm. Of the 73 randomized participants, 5 participants, 2 in the high dose and 3 in the low dose arms were randomized but did not receive surgery and did not take part in the study. 68 participants had surgery.
  For participants randomized to treatment dose, one eye was randomized to surgery and the fellow eye was randomized to sham.
Units Other Than Participants: eyes
Groups:
- Participants That Received Low Dose NT-501 Implant Surgery and Sham Surgery in Fellow Eye: NT-501 Low Dose Implant: encapsulated cell therapy that delivers ciliary neurotrophic factor to the retina
  Sham Surgery in Fellow Eye
- Sham Treatment in Fellow Eye for Low Dose Arm; Sham Treatment in Fellow Eye for High Dose Implant Arm: Sham Surgery in Fellow Eye for NT-501 Low Dose Implant Arm
- Participants That Received High Dose NT-501 Implant Surgery and Sham Surgery in Fellow Eye: NT-501 High Dose Implant: encapsulated cell therapy that delivers ciliary neurotrophic factor to the retina
  Sham Surgery in Fellow Eye
Period: Overall Study
Arm/Group | Participants That Received Low Dose NT-501 Implant Surgery and Sham Surgery in Fellow Eye | Sham Treatment in Fellow Eye for Low Dose Arm | Participants That Received High Dose NT-501 Implant Surgery and Sham Surgery in Fellow Eye | Sham Treatment in Fellow Eye for High Dose Implant Arm
Started (Participants screened, deemed eligible, randomized to a study arm) | 23; 23 eyes | 23; 23 eyes | 50; 50 eyes | 50; 50 eyes
NT-501 Surgery Completed | 20; 20 eyes | 20; 20 eyes | 48; 48 eyes | 48; 48 eyes
Completed (Study completion) | 18; 18 eyes | 18; 18 eyes | 44; 44 eyes | 44; 44 eyes
Not Completed | 5; 5 eyes | 5; 5 eyes | 6; 6 eyes | 6; 6 eyes
Not completed — Withdrawal by Subject | 1 | 1 | 4 | 4
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0
Not completed — Did not proceed with surgery | 3 | 3 | 2 | 2

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all 73 participants who were randomized to a treatment arm including the 3 participants from low dose arm and the 2 participants from the high dose arm who discontinued prior to surgery, and study start.
Units Other Than Participants: Eyes
Groups:
- Low Dose - Implant: NT-501 Low Dose Implant: encapsulated cell therapy that delivers ciliary neurotrophic factor to the retina
- Low Dose - Sham: Sham Implant in Fellow Eye (Low Dose Arm)
- High Dose - Implant: NT-501 High Dose Implant: encapsulated cell therapy that delivers ciliary neurotrophic factor to the retina
- High Dose - Sham: Sham Implant in Fellow Eye (High Dose Arm)
- Total: Total of all reporting groups
Arm/Group | Low Dose - Implant | Low Dose - Sham | High Dose - Implant | High Dose - Sham | Total
Number analyzed (Participants) | 23 | 23 | 50 | 50 | 73
Number analyzed (Eyes) | 23 | 23 | 50 | 50 | 146
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.9 (12.0) | 34.9 (12.0) | 40.2 (11.8) | 40.2 (11.8) | 37.6 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 26 | 26 | 74
  Male | 12 | 12 | 24 | 24 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 4 | 4 | 10
  Not Hispanic or Latino | 22 | 22 | 46 | 46 | 136
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 2
  Asian | 1 | 1 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 21 | 21 | 49 | 49 | 140
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Ocular History - Years Since RP Diagnosis [Mean (Standard Deviation); unit: years] | 8.85 (8.39) | 8.85 (8.39) | 10.49 (9.86) | 10.49 (9.86) | 10.00 (9.41)
Type of Ocular History [Number; unit: Eyes]
  Ocular disease | 23 | 23 | 50 | 50 | 146
  Ocular surgery | 3 | 3 | 10 | 11 | 27
  Ocular treatment | 0 | 0 | 2 | 4 | 6
Humphrey Visual Fields - Total Sensitivity (MITT Population) [Mean (Standard Deviation); unit: dB] — Humphrey Visual Field Sensitivity (VFS) is based on the HVF 30-2 test, consisting of 76 points; response measure was the sum of actual thresholds for all 76 locations, in dB (decibels). Foveal sensitivity was not used in assessing total. Population: MITT Population who received an implant
  dB
    number analyzed (Participants) | 20 | 20 | 48 | 48 | 68
    (all) | 1142.4 (446.33) | 1135.9 (423.50) | 969.8 (391.74) | 961.7 (435.68) | 1052.5 (424.31)

OUTCOME MEASURES:

1. Primary Outcome: Change in Humphrey Visual Fields - Total Sensitivity
Description: The primary efficacy endpoint was the change in Humphrey VFS from baseline to month 12 (Visit 10) as determined by the HVF 30-2 test, comprised of 76 points. The measure was the sum of actual thresholds for all 76 locations.
Time Frame: 12 months
Population: MITT Population excluding 1 participant from the high dose arm who did not complete any visits subsequent to surgery.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Low Dose - Implant | Low Dose - Sham | High Dose - Implant | High Dose - Sham
Number analyzed (Participants) | 20 | 20 | 47 | 47
dB | 1.4 (174.58) | 16.8 (165.41) | -164.8 (115.02) | -66.7 (103.23)

2. Secondary Outcome: Change in Mean Humphrey Visual Fields Sensitivity
Time Frame: Baseline compared to 6, 12, 18, 24 and 30 months
Population: MITT Population excluding 1 participant from the high dose arm who did not complete any visits subsequent to surgery.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Low Dose - Implant | Low Dose - Sham | High Dose - Implant | High Dose - Sham
Number analyzed (Participants) | 20 | 20 | 47 | 47
dB
  6 Months - Change from BL | -1.21 (140.09) | 25.80 (128.34) | -135.23 (107.86) | -42.99 (82.85)
  12 Months - Change from BL | 1.35 (174.58) | 16.75 (165.41) | -164.79 (115.02) | -66.65 (103.23)
  18 Months - Change from BL: number analyzed (Participants) | 20 | 20 | 46 | 46
  18 Months - Change from BL | -62.65 (208.64) | -37.33 (173.46) | -202.31 (137.13) | -98.73 (127.09)
  24 Months - Change from BL | -104.15 (194.50) | -72.15 (162.72) | -227.89 (149.73) | -136.96 (126.73)
  30 Months (retained implant) - Change from BL: number analyzed (Participants) | 12 | 12 | 25 | 25
  30 Months (retained implant) - Change from BL | -46.977 (345.78) | -58.64 (275.09) | -321.72 (196.81) | -211.82 (145.25)
  30 Months (6 Months Post-Explant) - Change from BL: number analyzed (Participants) | 6 | 6 | 20 | 20
  30 Months (6 Months Post-Explant) - Change from BL | -82.67 (185.60) | -58.50 (148.57) | -188.64 (122.33) | -144.60 (134.31)

3. Secondary Outcome: Mean Humphrey Visual Fields Sensitivity
Description: Change in Humphrey Visual Field Sensitivity over time
Time Frame: Baseline compared to 6, 12, 18, 24 and 30 months
Population: MITT Population
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Low Dose - Implant | Low Dose - Sham | High Dose - Implant | High Dose - Sham
Number analyzed (Participants) | 20 | 20 | 48 | 48
dB
  Baseline | 1142.43 (446.33) | 1135.94 (423.50) | 969.83 (391.74) | 961.70 (435.68)
  6 Months: number analyzed (Participants) | 20 | 20 | 47 | 47
  6 Months | 1141.21 (438.07) | 1161.74 (399.67) | 834.60 (354.98) | 918.72 (422.60)
  12 Months: number analyzed (Participants) | 20 | 20 | 47 | 47
  12 Months | 1143.78 (409.76) | 1152.69 (388.30) | 805.03 (357.86) | 895.05 (427.12)
  18 Months: number analyzed (Participants) | 20 | 20 | 46 | 46
  18 Months | 1079.78 (440.81) | 1098.61 (427.23) | 757.80 (363.86) | 850.92 (404.91)
  24 Months: number analyzed (Participants) | 20 | 20 | 47 | 47
  24 Months | 1038.28 (430.12) | 1063.79 (398.68) | 745.62 (344.58) | 825.06 (396.47)
  30 Months with retained implant: number analyzed (Participants) | 12 | 12 | 25 | 25
  30 Months with retained implant | 1176.22 (384.29) | 1173.32 (340.09) | 695.97 (251.57) | 787.30 (322.72)
  30 Months (6 Months Post-Explant): number analyzed (Participants) | 6 | 6 | 20 | 20
  30 Months (6 Months Post-Explant) | 1090.92 (382.10) | 1056.08 (406.65) | 752.78 (345.78) | 782.60 (382.68)

ADVERSE EVENTS:
Time Frame: Time of consent through Month 30 (study exit)
Description: Adverse events were followed from time of initial consent through 30 Months (study exit).
Arm/Group | Low Dose | High Dose
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/48
Serious Adverse Events (participants affected / at risk) | 1/20 | 4/48
Other Adverse Events (participants affected / at risk) | 20/20 | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=20) | High Dose (N=48)
Cubital tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Acute appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hypertrophic medial synovial plica with synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — right knee
Non-ischemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=20) | High Dose (N=48)
Anterior Chamber Cell (Eye disorders) | 7 (7) | 9 (9)
Anterior Chamber Flare (Eye disorders) | 5 (5) | 9 (9)
Asthenopia (Eye disorders) | 2 (2) | 1 (1)
Cataract Subcapsular (Eye disorders) | 1 (1) | 2 (2)
Conjunctival Haemorrhage (Eye disorders) | 17 (17) | 38 (38)
Conjunctival Hyperaemia (Eye disorders) | 12 (12) | 17 (17)
Conjunctival Oedema (Eye disorders) | 3 (3) | 6 (6)
Dellen (Eye disorders) | 1 (1) | 3 (3)
Diplopia (Eye disorders) | 1 (1) | 4 (4)
Eye Discharge (Eye disorders) | 2 (2) | 2 (2)
Eye Inflammation (Eye disorders) | 2 (2) | 4 (4)
Eye Irritation (Eye disorders) | 5 (5) | 4 (4)
Eye Pain (Eye disorders) | 6 (6) | 12 (12)
Eye Pruritis (Eye disorders) | 1 (1) | 3 (3)
Eyelid Oedema (Eye disorders) | 2 (2) | 2 (2)
Foreign Body Sensation in Eyes (Eye disorders) | 3 (3) | 11 (11)
Hypotony of Eye (Eye disorders) | 1 (1) | 2 (2)
Macular Oedema (Eye disorders) | 1 (1) | 5 (5)
Maculopathy (Eye disorders) | 0 (0) | 6 (6)
Miosis (Eye disorders) | 0 (0) | 15 (15)
Ocular Hyperaemia (Eye disorders) | 1 (1) | 4 (4)
Photophobia (Eye disorders) | 2 (2) | 3 (3)
Photopsia (Eye disorders) | 0 (0) | 4 (4)
Pupils Unequal (Eye disorders) | 1 (1) | 8 (8)
Vision Blurred (Eye disorders) | 1 (1) | 6 (6)
Visual Acuity Reduced (Eye disorders) | 1 (1) | 7 (7)
Visual Disturbance (Eye disorders) | 0 (0) | 4 (4)
Vitreous Detachment (Eye disorders) | 1 (1) | 6 (6)
Vitreous Disorder (Eye disorders) | 5 (5) | 7 (7)
Vitreous Floaters (Eye disorders) | 1 (1) | 4 (4)
Vitreous Haemorrhage (Eye disorders) | 1 (1) | 4 (4)
Vitreous Opacities (Eye disorders) | 1 (1) | 5 (5)
Implant Site Reaction (General disorders) | 0 (0) | 3 (3)
Influenza (Infections and infestations) | 1 (1) | 4 (4)
Nasopharyngitis (Infections and infestations) | 4 (4) | 9 (9)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 2 (2)
Corneal Abrasion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Periorbital Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Post Procedural Complication (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Post Procedural Discomfort (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Procedural Pain (Injury, poisoning and procedural complications) | 4 (4) | 6 (6)
Suture Related Complication (Injury, poisoning and procedural complications) | 5 (5) | 14 (14)
Intraocular Pressure Decreased (Investigations) | 1 (1) | 6 (6)
Intraocular Pressure Increased (Investigations) | 1 (1) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 5 (5) | 3 (3)
Depression (Psychiatric disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes